CLINICAL TRIAL: NCT04239898
Title: Feasibility, Acceptability, Tolerability, and Potential Health Effects of Microgreen Consumption in Healthy Middle-Aged and Older Adults
Brief Title: Microgreen Consumption for Healthy Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MG2019
Record Dates: First submitted 2019-11-12; First posted 2020-01-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aging; Menopause; Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red cabbage microgreens (Experimental): 2 cups of fresh red cabbage microgreens per day
  Interventions: Other: Red cabbage microgreens
- Red beet microgreens (Experimental): 2 cups of fresh red beet microgreens per day
  Interventions: Other: Red beet microgreens

INTERVENTIONS:
Other: Red cabbage microgreens — 2 cups per day
  Arms: Red cabbage microgreens
Other: Red beet microgreens — 2 cups per day
  Arms: Red beet microgreens

SUMMARY:
Microgreens are an emerging horticultural food crop with potential to improve human health. Previous research suggests they have broad consumer acceptance and that the micronutrient and bioactive compound levels are higher than that of their mature counterparts. To date, no studies have explored the feasibility of microgreen consumption, gastrointestinal tolerance of microgreen consumption, or their potential health impacts in humans. Therefore, the overall goal of this study is to explore the feasibility and acceptability of daily microgreen consumption, gastrointestinal tolerability, and potential health impacts of red cabbage and red beet microgreens in healthy middle-aged/older men and postmenopausal women - a population inherently at risk for chronic disease, e.g. cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal
* Aged 45-70

Exclusion Criteria:

* Cardiovascular disease, hypertension, diabetes, neuropathy, thrombosis, cancer, gastrointestinal, kidney, liver, lung, or pancreatic disease
* Taking medication for high cholesterol, triglycerides, or blood sugar, or are taking testosterone medications
* Blood pressure ≥ 130/80 mm Hg, triglyceride levels > 200 mg/dL, low-density lipoprotein cholesterol levels ≥ 160 mg/dL, total cholesterol levels ≥ 240 mg/dL, and/or hemoglobin A1c ≥ 6.5%
* Weight change ≥ 3 kg (6.6 lb.) in the past 3 months prior to starting the study, are actively trying to lose weight, or are unwilling to remain weight stable throughout the study
* Have a BMI less than 18.5 or greater than 30 kg/m2
* Are not willing to maintain normal eating/drinking and exercise habits over the duration of the study
* Currently smoke cigarettes or have a history of smoking cigarettes in the past 12 months
* Taking antibiotics or have taken them within one month of starting the study
* Binge and/or heavy drinker (>4 drinks on any given occasion and/or >14 drinks/week for men)
* Have allergies or contraindication to study foods, procedures, or procedure supplies

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants retained | Baseline to 6 weeks
  The number of participants retained versus lost to follow-up throughout the entire study
Adherence to the intervention | Baseline to 2 weeks
  Adherence will be determined for each 2-week microgreen intervention through a daily microgreen consumption log

SECONDARY OUTCOMES:
Gastrointestinal symptom self-assessment | Baseline to 2 weeks
  Determine the effects on gastrointestinal symptoms using a validated questionnaire for each 2-week microgreen intervention
Gastrointestinal health | Baseline to 2 weeks
  Determine the effects on gastrointestinal health using a daily bowel movement log for each 2-week microgreen intervention
Blood pressure | Baseline to 2 weeks
  Determine the effects on brachial and aortic blood pressure measured by SphygmoCor for each 2-week microgreen intervention
Augmentation index | Baseline to 2 weeks
  Determine the effects on augmentation index measured by SphygmoCor for each 2-week microgreen intervention
Microbiota modulation | Baseline to 2 weeks
  Use of 16s rRNA sequencing of stool samples to determine the effects of each 2-week microgreen intervention on microbial populations
Acceptability | 2-week visit
  Determine acceptability and feasibility of daily microgreen consumption through qualitative interviews with study participants at completion of the 2-week study

OTHER OUTCOMES:
Changes in plasma metabolites | Baseline to 2 weeks
  Use of mass spectrometry to determine the effects on plasma metabolites of bioactive compounds for each 2-week microgreen intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Science and Human Nutrition, Colorado State University, Fort Collins, Colorado, United States